CLINICAL TRIAL: NCT06050148
Title: Faecal Microbiota Transplantation as Means of Preventing Recurrent Urinary Tract Infections
Acronym: FMT-UTI
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Anu Kantele, Professor of infectious diseases, University of Helsinki and Helsinki University Hospital, Department of infectious diseases, Meilahti Vaccine Research Center MeVac, Helsinki, Finland, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMT-UTI
Record Dates: First submitted 2023-08-29; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: Urinary tract infection, Faecal microbiota transplantation, ESBL, Antimicrobial resistance; Recurrent urinary tract infection; UTI
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Part A: Double-blinded randomised trial for volunteers with recurrent UTIs with 1:1 FMT and placebo (PT) arms undergoing transfer of feces or placebo, respectively (Groups 1 and 2). Randomisation with respect to ESBL positivity (equal numbers of ESBL-positive in FMT and PT arms) and menopause. The groups will undergo an intensive 12-month follow-up.
  (Part B: a concomitant separate non-randomised follow-up study for non-trial participants, recruited separately, groups 3 and 4, no further description)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Unblinded team takes care of fecal microbiota transplantion but does not participate in other parts of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feacal microbial transplantation (FMT) (Experimental)
  Interventions: Biological: Feacal microbial transplantation (FMT)
- Placebo transplantation (PT), transplantation with coloured 0,9% NaCl-solution (Placebo Comparator)
  Interventions: Other: Placebo transplantation (PT)

INTERVENTIONS:
Biological: Feacal microbial transplantation (FMT) — Feacal microbial transplantation (FMT)
  Arms: Feacal microbial transplantation (FMT)
Other: Placebo transplantation (PT) — Transplantation with coloured 0,9% NaCl-solution
  Arms: Placebo transplantation (PT), transplantation with coloured 0,9% NaCl-solution

SUMMARY:
This study investigates Faecal microbiota transplantation (FMT) in prevention of recurrent urinary tract infections (UTIs) caused either by sensitive E. coli or ESBL-E. coli.

ELIGIBILITY:
Inclusion criteria:

* Female subjects aged ≥18
* History of recurrent UTI: at least two episodes of UTI over the past 6 months or at least three episodes over the past year, most recent episode within the past three months
* Written informed consent

Exclusion criteria:

* Suspected non-compliance
* Diagnosis of a gastrointestinal disease
* Pregnancy
* Immunosuppression
* Any kind of permanent urinary catheter or intermittent urinary catheterization
* Any other criteria which, in the investigator's opinion, would compromise the ability of the subject to participate in the study, the subject's well-being, or the outcome of the study

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
mean number of UTI episodes after FMT among patients with recurrent UTI | 12 months
proportion of participants with UTI after FMT among patients with recurrent UTI | 12 months

SECONDARY OUTCOMES:
mean number of UTI episodes caused by sensitive E. colis after FMT among patients with recent non-ESBL/MDR UTIs | 12 months
proportion of participants with UTIs caused by sensitive E. colis after FMT among patients with recent non-ESBL/MDR UTIs | 12 months
mean number of UTI episodes caused by ESBL/MDR E. colis after FMT among patients with recent ESBL/MDR UTIs | 12 months
proportion of participants with UTIs caused by ESBL/MDR E. colis after FMT among patients with recent ESBL/MDR UTIs | 12 months
identifying groups of bacteria associated with smaller number of UTI episodes after FMT | 12 months
the duration of successful prevention by FMT | 1-5 years
proportion of participants with recurrent UTI and concurrent intestinal MDR colonisation with the same strain | 12 months
proportion of participants with intestinal ESBL/MDR eradicated after FMT | 1-12 months
confirm whether the uropathogen are identical before and after FMT | 12 months
  evaluated by antimicrobial sensitivity profile and whole-genome sequencing
number of antibiotic courses received by FMT versus placebo recipients | 12 months
proportion of participants with gastrointestinal symptoms assessed by GSRS scores before and after FMT | 1-12 months
  Gastrointestinal symptom rating scale -questionnaire with 15 items on a 7-level Likert scale (1-7), higher scores for more intense symptoms during the past week
proportion of participants with mild to severe depression assessed by BDI scores before and after FMT | 1-12 months
  Beck's Depression Inventory: 21-question multiple-choice self-report inventory, higher scores for more severe depression
mean number of health-related quality of life (HRQoL) scores assessed by 15D before and after FMT | 1-12 months
  Quality of life -questionnaire (15D): a generic, comprehensive (15-dimensional), self-administered questionnaire, lower scores for better HRQoL
description of groups of bacteria in faecal and urine microbiome before and after FMT | 12 months
human urine and serum metabolic profiles before and after FMT | 12 months
  assessed by a 1H-Nuclear Magnetic Resonance-based metabolomic approach

CONTACTS AND LOCATIONS:
Locations (1):
- Meilahti Vaccine Research Center, Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: HUS informational website for recruitment — https://www.hus.fi/ulosteensiirto-toistuvien-virtsatieinfektioiden-ehkaisyssa-tule-mukaan-tutkimukseen